CLINICAL TRIAL: NCT00185978
Title: School- and Family-Based Obesity Prevention for Children
Brief Title: Obesity Prevention for Pre-Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HL054102 (NIH); R01HL054102 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
Keywords: obesity prevention; preadolescents; schools
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity | interventions — Diet; Exercise

INTERVENTIONS:
Behavioral: diet, physical activity, reduced sedentary behavior

SUMMARY:
To develop and evaluate, in a randomized controlled trial, a comprehensive obesity prevention program for third, fourth and fifth grade students.

The intervention includes activities in THE SCHOOL, THE HOME, and a clinically oriented component for HIGH-RISK CHILDREN. In addition, the intervention will be delivered over a 3 year period, with age and grade-appropriate components for 3rd, 4th and 5th graders and their families. The primary outcome is body mass index.

PRIMARY OBJECTIVE: To significantly reduce body mass index, compared to controls, at the end of the three year intervention.

DETAILED DESCRIPTION:
To develop and evaluate, in a randomized, controlled trial, a comprehensive obesity prevention program for third, fourth and fifth grade students.

Late childhood and early adolescence appears to be an important period in the development of obesity. Physiologic changes associated with puberty may increase the risk of acquiring clinically significant obesity. Onset of obesity in early adolescence appears to be associated with increased risks of "tracking" of obesity into adulthood, obesity-associated morbidity and mortality in adulthood, and obesity-associated psychosocial morbidity. However, (1) we have a limited ability to accurately identify those children who will become obese adults and those who will suffer obesity-related morbidities, (2) most existing treatments for overweight children and adolescents have yielded modest, unsustained effects, and (3) single-component preventive interventions have been relatively ineffective. Acknowledging these observations, the consensus at the recent NHLBI Strategy Development Workshop for Public Education on Weight and Obesity was that population-based primary and secondary prevention efforts, targeting pre-adolescents, may hold the greatest promise for addressing the problem of obesity. Therefore, we propose an integrated, multiple-component, school and family-based, primary and secondary prevention program targeting third, fourth and fifth graders.

Our proposed intervention model is derived directly from principles of Bandura's social cognitive theory. The intervention includes activities in THE SCHOOL, THE HOME, and a clinically oriented component for HIGH-RISK CHILDREN. In addition, the intervention will be delivered over a 3 year period, with age and grade-appropriate components for 3rd, 4th and 5th graders and their families.

We will evaluate the efficacy of our comprehensive intervention in a cohort of third graders, in ethnically diverse elementary schools. Schools will be randomly assigned to the comprehensive intervention or an attention-placebo curriculum, to minimize the potential for compensatory rivalry or resentful demoralization. Assessments of children's height, weight, triceps skinfold thickness, waist and hip circumferences, food preferences, cardio-respiratory fitness, and self-reported behavior, attitudes, and knowledge will occur every 6 months, and 6-months following the end of the intervention. The primary outcome is body mass index.

PRIMARY OBJECTIVE: To significantly reduce body mass index, compared to controls, at the end of the three year intervention.

ELIGIBILITY:
Inclusion Criteria:

* all third graders in the participating elementary schools at baseline

Exclusion Criteria:

* unable to complete the study procedures

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Start 1998-04; Study Completion 2001-03

PRIMARY OUTCOMES:
body mass index

SECONDARY OUTCOMES:
prevalence/incidence of obesity
prevalence of obesity among high risk children
resting heart rate
moderate to vigorous physical activity
hours of television viewing
fat intake
preferences for low fat, high fiber foods
weight concerns
knowledge and attitudes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N. Robinson, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Robinson TN, Killen JD. Obesity prevention for children and adolescents. In: Thompson, J.K., & Smolak, L. (Eds.) Body Image, Eating Disorders, and Obesity in Youth: Assessment, Prevention, and Treatment. Washington, DC: American Psychological Association, 2001, pp. 261-292.